CLINICAL TRIAL: NCT01505543
Title: Proprioceptive Postural Control and Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Simon Brumagne, Prof. dr. Simon Brumagne, KU Leuven
Other Study IDs: 2012_SBrumagne_COPD; 1.5.104.03, G.0674.09 (Other Grant/Funding Number: Research Foundation Flanders (FWO))
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2012-07

CONDITIONS: Proprioceptive Postural Control; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- chronic obstructive pulmonary disease
- healthy matched controls

SUMMARY:
Proprioceptive weighting changes may explain differences in postural control performance. In addition, the respiratory movement has a disturbing effect on postural balance. Postural balance seems to be impaired in individuals with respiratory disorders. Increased risk of falling is reported in individuals with chronic obstructive pulmonary disease. Besides the essential role of respiration, the diaphragm may also play an important role in the control of the trunk and postural balance.

The aim of the study is to clarify whether proprioceptive postural control is impaired in individuals with chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria individuals with chronic obstructive pulmonary disease:

* Age: 40-80 years old
* Spirometry (post-bronchodilator) based diagnosis of COPD (GOLD criteria)
* Willingness to sign the informed consent

Inclusion Criteria healthy controls:

* Age: 40-80 years old
* No COPD (spirometry based: FEV1/FVC ≥ 0.7 and FEV1 > 80%)
* Willingness to sign the informed consent

Exclusion Criteria:

* History of major trauma and/or major orthopedic surgery of the spine, the pelvis or the lower quadrant
* One of the following conditions: Parkinson, multiple sclerosis, stroke, history of vestibular disorder
* Respiratory disorder other than COPD
* α1-antitrypsin deficiency
* Known history of significant inflammatory disease other than COPD
* COPD exacerbation within 4 weeks prior to study
* Lung surgery
* Recent diagnosis of cancer
* Therapy with oral corticosteroids in the last 6 weeks
* Significant cardiovascular comorbidity

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients from the University Hospital Leuven - Respiratory Disvision
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Proprioceptive postural control | 6 months
  Center of pressure displacement (force plate) in standing in response to local muscle vibration on ankle and back muscles to specifically detect the role of proprioception in postural control.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Brumagne, PhD, Principal Investigator — KU Leuven; Thierry Troosters, PhD, Principal Investigator — KU Leuven; Wim Janssens, MD, PhD, Principal Investigator — KU Leuven; Marc Decramer, MD, PhD, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Janssens L, Brumagne S, Polspoel K, Troosters T, McConnell A. The effect of inspiratory muscles fatigue on postural control in people with and without recurrent low back pain. Spine (Phila Pa 1976). 2010 May 1;35(10):1088-94. doi: 10.1097/BRS.0b013e3181bee5c3. PMID 20393397